CLINICAL TRIAL: NCT01360463
Title: Efficacy of Drug-HIV Counseling Among IDU at Methadone Clinics in Jakarta
Brief Title: Efficacy of Drug and Risk Counseling Among Methadone Patients in Jakarta, Indonesia
Acronym: JAKPRO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: David S. Metzger, Ph.D. , Principal Investigator, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JAKPRO; R01DA026344 (NIH)
Record Dates: First submitted 2011-05-23; First posted 2011-05-25 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2011-05

CONDITIONS: HIV Risk Behaviors; Heroin Injection; Retention in Methadone Treatment
Keywords: drug abuse counseling; HIV risk reduction counseling; HIV infection; injection drug users; AIDS
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Behavioral and Drug Risk Counseling (Experimental): Participants assigned to this arm will receive bi weekly Behavioral and Drug Risk Counseling (BDRC) counseling for six months.
  Interventions: Behavioral: Behavioral Drug and Risk Counseling (BDRC)
- Treatment as Usual (Active Comparator): Participants assigned to this arm will receive methadone treatment without and alterations.
  Interventions: Behavioral: methadone maintenance treatment

INTERVENTIONS:
Behavioral: Behavioral Drug and Risk Counseling (BDRC) — The BDRC counseling is rooted in cognitive behavioral theory. During one hour sessions, the counselors help participant identify short term behavioral goals and work with the participant to develop strategies to achieve their goals. These plans are referred to as "contracts" and these contracts are reviewed and revised at each subsequent session.
  Arms: Behavioral and Drug Risk Counseling
Behavioral: methadone maintenance treatment — daily individualized doses of methadone will be provided by the program staff.
  Arms: Treatment as Usual

SUMMARY:
According to UNAIDS, Indonesia is experiencing one of the most rapidly expanding HIV/AIDS epidemics in Asia. The epidemic in Indonesia has been fueled by injection drug use among heroin users and the national response includes the scale-up of methadone maintenance treatment.

Drug counseling is considered to be an integral part of methadone treatment, but few studies have been designed to assess its benefits and costs. In settings such as Jakarta, data regarding the costs and benefits of drug counseling have critical public heath relevance.

The investigators propose to conduct a prospective randomized trial to evaluate the efficacy of integrated drug and HIV counseling among injecting drug users. This study will be conducted at six methadone clinics in Jakarta, Indonesia where the HIV prevalence among injecting drug users ranges between 50- 86%, with collaborators from the Drug Dependence Hospital in Jakarta, the University of Pennsylvania and Yale University. The specific aims of this four year study are to evaluate the impact of Behavioral Drug and Risk Counseling (BDRC)-a low intensity, cognitive behavioral approach that integrates drug counseling and risk reduction intervention. Those assigned to the BDRC arm will be compared to those who receive treatment as usual which includes an initial risk reduction intervention and counseling as needed. The investigators hypothesize that the structured, low intensity BDRC approach will be more cost effective and result in higher rates of retention in treatment, lower rates of drug use and lower rates of HIV risk.

To test these hypotheses, the research team in Jakarta will recruit 300 injecting drug users as they enter treatment at the Drug Dependence Hospital and its five satellite programs. Following informed consent procedures, research staff will randomize participants to either the BDRC intervention or to treatment as usual. All subjects will be fuly assessed at baseline and months 3, 6, 9, and 12.

The proposed work will be build on collaborations that have been established with the Indonesian Investigator Adhi Nurhidayat,MD during his NIDA INVEST Fellowship at University of Pennsylvania when he spent time with David Metzger, PhD and George Woody, MD. It will also extend findings from a WHO study on substitution therapy of opiates and HIV/AIDS that was completed by Riza Sarasvita, MS,MHS (former NIDA Humphrey Fellow at Johns Hopkins University) and her colleagues at The Drug Dependence Hospital Jakarta, Indonesia.

ELIGIBILITY:
Inclusion Criteria:

* Enrollment in methadone maintenance treatment
* Injected heroin within past 30 days by self-report, documented by "tracks" or puncture marks
* 18 or more years of age
* Meets DSM-IV criteria for opiates dependence with physiologic features
* Agrees to keep bi-weekly appointments if selected
* Current address within Jakarta and not planning to move
* Willingness and ability to give informed consent and otherwise participate
* Provision of adequate locator information

Exclusion Criteria:

* Clinically significant cognitive impairment, schizophrenia, paranoid disorder, bipolar disorder
* Advanced neurological, cardiovascular, renal, or other medical disorder that is likely to impair or make hazardous patient's ability to participate
* Physiologically dependent on alcohol, benzodiazepines or other sedative type drugs
* Concurrent participation in another treatment study
* Planning to enter inpatient or residential treatment within next year
* Pending legal charges with likely incarceration within next 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 276 (Actual)
Dates: Start 2009-05; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Injection drug use | one year
  the primary endpoint will be the frequency of injection drug use during the 30 days prior to the final assessment at 12 months.

SECONDARY OUTCOMES:
retention in methadone treatment | one year
  number of months retained in treatment during the one year assessment period.

CONTACTS AND LOCATIONS:
Locations (1):
- RSKO Drug Dependence Hospital, Jakarta, Timur, Indonesia